CLINICAL TRIAL: NCT04435340
Title: Clinical and Sonographic Outcome After Ventral Abdominal Hernia Repair With Self Adhering, Atraumatic Mesh in the Retro-rectus (Sublay) Position
Brief Title: Ventral Abdominal Hernia Repair With Self Adhering, Atraumatic Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spital Limmattal Schlieren (Other)
Responsible Party: Principal Investigator, Prof Urs Zingg, Head of Department of Surgery, Spital Limmattal Schlieren
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018-00122
Record Dates: First submitted 2020-01-07; First posted 2020-06-17 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Abdominal Hernia
Keywords: Abdominal Hernia; Ventral Hernia; Atraumatic mesh
MeSH Terms: conditions — Hernia, Abdominal; Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: retro- and prospective arm
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective (Other): All patients in the retrospective cohort are contacted at least 1 year after surgery and/or 3 years after surgery via phone call or letter, informed about the study and asked to participate. In case of informed consent, they are invited to the study site. They are asked to complete the questionnaires and they undergo a Sonography of the ventral abdomen.
  Interventions: Diagnostic Test: Selective Sonography of the ventral abdominal hernia level
- Prospective (Other): All patients in the prospective cohort are informed about the study and asked to participate in the outpatient clinic before surgery. In case of informed consent, they are invited to the study site at least one year and three years, respectively, after surgery. They are asked to complete the questionnaires and they undergo an ultrasound of the ventral abdomen.
  Interventions: Diagnostic Test: Selective Sonography of the ventral abdominal hernia level

INTERVENTIONS:
Diagnostic Test: Selective Sonography of the ventral abdominal hernia level — The primary outcome of the study is measured by an radiologist experienced in abdominal ultrasound with a linear ultrasound transducer (ML 6-15 Hz). In case of aggravated examination circumstances a different ultrasound transducer is used (linear 9 L or convex C 1-6 Hz)

SUMMARY:
Patients who underwent ventral abdominal hernia repair with self adhering, atraumatic mesh in sublay position are examined for their recurrence rate

DETAILED DESCRIPTION:
The study includes all patients operated from 11.03.2014 to 31.12.2020. Patients will undergo a Sonography at least one year after surgery. The patients operated form 11.03.2014 to date are therefore a retrospective cohort, the patients from to date until 31.12.2020 a prospective cohort. This method is used to achieve the highest possible number of patients in a define period of time with no alteration of surgical technique.

All patients in the retrospective cohort are contacted at least 1 year after surgery and/or 3 years after surg ery via phone call or letter, informed about the study and asked to participate. In case of informed consent, they are invited to the study site. They are asked to complete the questionnaires and they undergo a Sonography of the ventral abdomen.

All patients in the prospective cohort are informed about the study and asked to participate in the outpatient clinic before surgery. In case of informed consent, they are invited to the study site at least one year and three years, respectively, after surgery. They are asked to complete the questionnaires and they undergo an ultrasound of the ventral abdomen.

The latest follow up should be completed by 31.03.2022.

For both, the retro- and prospective arm, the time needed for the follow-up appointment is approximately 1 hour. The completion of the ultrasound is estimated to take 20 minutes, the questionnaires is estimated to take 20-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Initially suffering from ventral abdominal hernia
* Performance of open ventral abdominal hernia repair with self-adhering, atraumatic mesh (Adhesix ®)
* Informed Consent as documented by signature (Appendix: Informed Consent Form)

Exclusion Criteria:

* Inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrance rate in sonography | 12 months after surgery
  The primary outcome is the recurrence rate of ventral abdominal hernia determined by clinical examination and sonography. A recurrence is defined if intraabdominal structures (i.e. intestines, omentum, preperitoneal fat tissue) reach ventrally of the facial layers .
Recurrance rate clinically | 12 months after surgery
  The primary outcome is the recurrence rate of ventral abdominal hernia determined by clinical examination. A recurrence is defined if intraabdominal structures (i.e. intestines, omentum, preperitoneal fat tissue) reach ventrally of the facial layers .

SECONDARY OUTCOMES:
Pain and sensation of the mesh measured by the Carolinas Comfort Scale questionnaire | 12 months after surgery
  Clinical subjective outcome 1
Limitations in quality of life questionnaire | 12 months after surgery
  Clinical subjective outcome 2
Daily activities measured HerQLes questionnaire | 12 months after surgery
  Clinical subjective outcome 3

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, Study Chair — Spital Limmattal Schlieren
Locations (1):
- Spital Limmattal, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No